CLINICAL TRIAL: NCT05465356
Title: Patient Engagement With Digital Health Tools in Rheumatology
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Nikita Arumalla, Principal investigator, Guy's and St Thomas' NHS Foundation Trust
Other Study IDs: EDGE 147423
Record Dates: First submitted 2022-06-22; First posted 2022-07-19 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Rheumatic Disease; PROM
Keywords: digital tools
MeSH Terms: conditions — Rheumatic Diseases | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- New patients: All new referrals seen in the rheumatology outpatients department, completing pre-appointment digital questionnaires
  Interventions: Other: Questionnaire; Other: Semi-structured interview
- Follow-up patients: Patient with inflammatory arthritis completing ePROMs [electronic Patient Reported Outcome Measures] through the remote monitoring platform
  Interventions: Other: Questionnaire; Other: Semi-structured interview

INTERVENTIONS:
Other: Questionnaire — Questionnaires completed as part of routine care - this is an observational study
Other: Semi-structured interview — Semi-structured interview to review factors involved in patients engaging or not-engaging with the digital tools

SUMMARY:
The purpose of this study is to evaluate the patient engagement with digital tools for diagnosis and monitoring of disease in rheumatology services

DETAILED DESCRIPTION:
The investigators plan to undertake a mixed methods study to investigate a digital algorithm to potentially inform triage of new patient referral to rheumatology services, as well as to inform follow up review schedules. Current practice at out hospital is to ask all newly referred patients to complete a pre-appointment digital questionnaire prior to their clinic visit. Patients who need follow up are then routinely invited to continue to return interval questionnaires related to their symptoms between clinic visits.

The investigators believe that the questionnaire responses could enable appropriate (and safe) allocation to a particular clinic (e.g. urgent early arthritis clinic or general rheumatology clinic for a new referral), or define an appropriate clinic follow up interval for a repeat visit for patients with a rheumatic disease.

Our study aims to evaluate these questionnaires using data collected from routine clinical practice, as well a series of semi-structured interviews with service users.

ELIGIBILITY:
Inclusion Criteria: quantitative phase:

* Aged 18 years and above
* Able to complete the questionnaire in English

  1. New patient pre-appointment questionnaires
* Referred as a new patient to the rheumatology outpatient department at Guys and St Thomas' Trust between 01/01/2019 to 01/10/2023 and sent a digital pre-appointment questionnaire
* Electronic patient notes recorded between 01/01/2019 to 01/10/2024

  2. Follow up patients PROM questionnaires
* Patients under followup of the rheumatology department at Guys and St Thomas' Trust with a diagnosis of rheumatoid arthritis, psoriatic arthritis or axial spondyloarthropathy who have been added to the remote monitoring program between 01/01/2019 to 01/10/2023
* Electronic patient notes recorded between 01/01/2019 to 01/10/2024

Inclusion criteria: qualitative phase:

* Aged 18 years and above

  1. New patient pre-appointment questionnaires
* Referred as a new patient to the rheumatology outpatient department at Guys and St Thomas' Trust between 01/01/2019 to 01/10/2023 and sent a digital pre-appointment questionnaire
* Able to communicate in English or any language offered for audio interpreting by the LanguageLine service

  2. Follow up patients PROM questionnaires
* Patients under followup of the rheumatology department at Guys and St Thomas' Trust with a diagnosis of rheumatoid arthritis, psoriatic arthritis or axial spondyloarthropathy who have been added to the remote monitoring program between 01/01/2019 to 01/10/2023
* Able to communicate in English or any language offered for audio interpreting by the LanguageLine service

Exclusion Criteria: quantitative phase:

* Under 18 years of age
* Unable to complete study questionnaires

Exclusion criteria: qualitative phase:

* Under 18 years of age
* Patients lacking the capacity to consent for themselves for the semi-structured interview

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All new patients referred to rheumatology outpatients + patients with inflammatory arthritis under follow up in rheumatology outpatients
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Number of patients with a non-inflammatory diagnosis | 3 years
  Clinician assessed diagnosis as categorised into inflammatory [e.g. rheumatoid arthritis] or non-inflammatory [e.g osteoarthritis or fibromyalgia]
Clinician assessed DAS-28 score for patients with rheumatoid arthritis | 3 years
  Clinician assessment of disease activity at next follow-up visit for remote monitoring questionnaires
Clinician assessed PsARC score for patients with psoriatic arthritis | 3 years
  Clinician assessment of disease activity at next follow-up visit for remote monitoring questionnaires
Rate of response to digital questionnaires | 3 years
  Proportion of patients completing the new patient pre-appointment and follow-up remote monitoring questionnaires.

SECONDARY OUTCOMES:
PHQ8 scores in new patients completing pre-appointment questionnaires | 3 years
  To estimate the prevalence of depression in new referrals to the rheumatology service. Score range 0 to 24, with higher score indicating more severe depression
GAD7 scores in new patients completing pre-appointment questionnaires | 3 years
  To estimate the prevalence of anxiety in new referrals to the rheumatology service. Score range 0 to 21, with higher score indicating more severe anxiety

CONTACTS AND LOCATIONS:
Overall Officials: Toby Garrood, FRCP, PhD, Study Chair — Guy's and St Thomas' NHS Foundation Trust

IPD SHARING:
Plan to Share IPD: No